CLINICAL TRIAL: NCT07235995
Title: Impact of Paracetamol and Mannitol Injection Analgesia on Postoperative Delirium in Elderly Patients After Non-cardical Surgery: A Randomized Controlled Trial
Brief Title: Paracetamol and Mannitol Injection and Postoperative Delirium
Acronym: PAPOD-ES
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, icuzhanglina, Professor, Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 202510115; 202510115 (Other: Xiangya Hospital)
Record Dates: First submitted 2025-11-13; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Delirium; Elderly; Non Cardiac Surgery
Keywords: Postoperative delirium; Intravenous acetaminophen; Elderly; Noncardiac surgical patients
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetaminophen group (Experimental): Intravenous acetaminophen is the analgesic of choice for patients in the acetaminophen group
  Interventions: Drug: Acetaminophen group
- Sufentanil group (Active Comparator): Intravenous sufentanil is the analgesic of choice for patients in the sufentanil group
  Interventions: Drug: Sufentanil group

INTERVENTIONS:
Drug: Acetaminophen group — The pain in this group is controlled using acetaminophen (Paracetamol and Maninitol Injection, Yichang Renfu Medicine Co., Ltd., China), 500 mg, intravenous bolus, every 6 hours for the first 48 hours postoperatively. The severity of pain is assessed using NRS every 15 minutes during the first hour following ICU admission and then once every 12 hours needed.
  Arms: Acetaminophen group
Drug: Sufentanil group — he pain in this group is controlled using sufentanil (Yichang Renfu Medicine Co., Ltd., China) intravenous infusion with a rate of 0.05 μg/kg/h. The severity of pain is assessed using NRS every 15 minutes during the first hour following ICU admission and then once every 12 hours needed.
  Arms: Sufentanil group

SUMMARY:
The aim of this multi-center RCT is to investigate the effect of intravenous acetaminophen (paracetamol and mannitol injection) on postoperative delirium, comparing with intravenous sufentanil, in elderly noncardiac surgical patients admitted to ICU.

DETAILED DESCRIPTION:
Delirium is a common complication after surgery. It is associated with increased morbidity and mortality, longer intensive care unit (ICU) and hospital stay, prolonged mechanical ventilation, higher risk of institutionalization, and higher healthcare cost. Depending on patient population and screening method, the incidence of delirium in elderly patients admitted to ICU can be as high as 58-76%. The choice of analgesics and the adequacy of pain control are among the modifiable precipitating factors for postoperative delirium (POD). Whether the use of intravenous acetaminophen decreases the occurrence of POD in elderly noncardiac surgical patients admitted to ICU remains inadequately studied.

Objectives: To investigate the effect of intravenous acetaminophen (paracetamol and mannitol injection) on postoperative delirium, comparing with intravenous sufentanil, in elderly noncardiac surgical patients admitted to ICU.

Study design: A randomized controlled trial. Setting: 34 ICUs from different regions across China. Patients: 1092 elderly patients (≥ 60 years), having noncardiac surgery and admitted to ICU after surgery, are eligible.

Intervention: Patients are randomly assigned to intravenous acetaminophen or sufentanil groups. Intravenous acetaminophen is the analgesic of choice for patients in the acetaminophen group. Intravenous sufentanil is the analgesic of choice for patients in the sufentanil group (control).

Outcomes: The primary endpoint is the incidence of delirium within the first 5 days after surgery. Delirium is assessed using the confusion assessment method for the intensive care unit (CAM-ICU). The secondary endpoints include the level of pain assessed using the Numeric Rating Scale (NRS) on postoperative day 1 to 5 and day 30, 30-day mortality, length of ICU and hospital stay, quality of life assessed on postoperative day 30, cognitive function assessed on postoperative day 30, and biomarkers and neurofunctional testing for delirium.

Predicted duration of the study: 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years;
* Admitted to ICU after a noncardiac surgical procedure
* Moderate to severe acute pain, with a postoperative pain score ≥ 5 based on the 11-point Numerical Pain Rating Scale (NPRS)
* Signed informed consent form

Exclusion Criteria:

* Preoperative medical history: schizophrenia, epilepsy, Parkinson's disease, or severe myasthenia gravis
* History of psychiatric disease or significant neurocognitive disorder such as dementia or retardation, making POD assessment impossible
* Language or communication barrier making POD assessment impossible
* Intracranial surgery
* Severe hepatic dysfunction prohibiting the use of acetaminophen per the standard of care
* Participation in a competing study within 30d
* Patients experienced intraoperative or postoperative complications, and the investigator determined the subject was unsuitable to continue participation in the study
* Intolerant to paracetamol or opioid drugs

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1092 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of delirium | postoperative 1- 5 days
  Delirium assessed using CAM-ICU every 12 hours (8am, 8 pm) during postoperative days 1-5 and RASS transform at any time

SECONDARY OUTCOMES:
All-cause mortality | 30-day after surgery
  30-days outcome (survival or death) after surgery; Patients will be assessed via phone call if they are discharged before day 30 after surgery
Severity of pain | postoperative days 1-5
  Severity of pain assessed using numeric rating scale (NRS), 8am and 8pm, twice a day, for 5 day The scale consists of 11 points from 0 to 10, where 0 indicates "no pain" and 10 indicates "severe pain". Patients select the corresponding number based on their pain level. <4 points indicate mild pain (no impact on sleep), 4-6 points indicate moderate pain, and ≥7 points indicate severe pain (pain prevents sleep or causes waking).
Length of ICU stay | immediately after surgery
  Length of ICU stay after surgery admitted to ICU
Length of hospital stay | immediately after surgery
  Length of hospital stay within hospital admission
Quality of life of 30-day survivors | day 30 after surgery
  Patients will be assessed with World Health Organization Quality of Life Assessment Instrument Short Form (WHOQOL-BREF) via phone call if they are discharged before day 30 after surgery The scale contains 26 items covering four domains: physiological, psychological, social relations, and environmental. It uses a 1-5-point Likert scale for scoring, and the original scores are converted into a standard score of 0-100. The higher the score, the better the quality of life.
Cognitive function of 30-day survivors | day 30 after surgery
  Patients will be assessed with TICS-m via phone call if they are discharged before day 30 after surgery
Incidence of non-delirium-related complications | 30 days after surgery
  Complications unrelated to delirium occurring within 30 days postoperatively (e.g., cardiovascular events, cerebrovascular events, renal impairment, GI complications, infections, etc.) are defined as any newly developed complications that may affect patient recovery and require therapeutic intervention (including hospital admission).

OTHER OUTCOMES:
Sleep quality | postoperative days 1-5
  Subjective quality of sleep assessed using NRS (an 11-point scale where 0 = the best sleep and 10 = the worst sleep) once daily (8:00-10:00 am) during postoperative days 1-5
Biomarker of delirium | Postoperative day 1
  Biomarker of delirium including S100b and NSE on postoperative day 1
Neuro monitoring of delirium | Postoperative days 1-5
  Monitoring of neurophysiological function, with detecting SctO2 during postoperative days 1-5

CONTACTS AND LOCATIONS:
Overall Officials: Yixiong Li, Study Chair — Central South University
Locations (1):
- Xiangya hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No